CLINICAL TRIAL: NCT04938960
Title: Identification of Non-gal, Non-HLA Antigens in Patients Implanted With Xenogenic Material
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Leigh G. Griffiths, Associate Professor of Medicine, Mayo Clinic
Other Study IDs: 17-007803
Record Dates: First submitted 2021-06-22; First posted 2021-06-25 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Valve Heart Disease
MeSH Terms: conditions — Heart Valve Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Biological Heart Valve: Participants receiving a biological heart valve
  Interventions: Diagnostic Test: blood draw
- Mechanical Heart Valve: Participants receiving a mechanical heart valve
  Interventions: Diagnostic Test: blood draw

INTERVENTIONS:
Diagnostic Test: blood draw — blood will be drawn at pre-operation, between 2 weeks and 3 months, between 3-11 months (optional; we will collect a sample if the patient returns to Mayo Clinic for any other non-study related visit), and between 12-18 months post-operatively.

SUMMARY:
This study involves collecting serum samples from patients presenting for aortic valve replacement at Mayo Clinic, Rochester, MN. Serum samples will be collected pre-op, between 2 weeks and 3 months, between 3-11 months (optional), and between 12-18 months post-operatively. The patients antibodies in these serum samples will be used to capture proteins from the same type of tissue their replacement heart valves are made from (i.e., bovine/porcine pericardium - a non-human tissue which is currently used to make glutaraldehyde-fixed heart valves). The captured proteins will be identified, and compared over time (i.e., 0, 1, 3 and 12 months) to determine which proteins (i.e., antigens) in bovine/porcine pericardium that the patient is mounting an immune response towards.

DETAILED DESCRIPTION:
Protein G HP SpinTrap columns will be used to capture IgG antibodies from patient serum pre-implant, between 2 weeks-3 months, between 3-11 months and between 12-18 months post-implant. These antibodies will be cross-linked to the column and then protein extracted from implant tissue (ie Native bovine/porcine pericardium) will be deglycosylated and run through the column. Antigenic proteins will be trapped and non-antigenic proteins will be washed through the column. These antigenic proteins will be eluted off the column and identified using LC-MS/MS. The proteins identified in the pre-implant elutant will be compared to the proteins in post-implant elutant to identify xenoantigens. Success criteria will be method validation by identification of previously known and new currently unknown xenoantigens.

ELIGIBILITY:
Inclusion Criteria:

* patients who will receive either a biological or mechanical heart valve

Exclusion Criteria:

* Currently receiving therapy for cancer requiring treatment with concurrent radiotherapy and/or chemotherapy
* Cancer in remission for less than 5 years if previously treated with radiotherapy and/or chemotherapy
* Previous tissue valve implants
* Current pregnancy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult males and females who will receive either a mechanical or biological heart valve implant
Sampling Method: Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Identify Non-gal, non-HLA protein antigens in patients that have received xenogenic tissue implant. | Approximately 12-18 months post-operatively
  The captured proteins will be identified, and compared over time (i.e., pre-op, between 2 weeks and 3 months, between 3-11 months (optional), and 12-18 months post-operatively) to determine which proteins (i.e., antigens) in bovine/porcine pericardium that the patient is mounting an immune response towards.

CONTACTS AND LOCATIONS:
Overall Officials: Leigh G Griffiths, PhD, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Mayo Clinic Florida, Jacksonville, Florida
  - Mayo Clinic Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No